CLINICAL TRIAL: NCT01659944
Title: A Single-site, Open-label, Fixed-sequence Phase 1 Study Evaluating the Effect of Eliglustat (Genz-112638) on the Pharmacokinetics, Safety and Tolerability of Metoprolol in Healthy Adult Subjects.
Brief Title: Study to Evaluate the Effect of Eliglustat on the Pharmacokinetics, Safety and Tolerability of Metoprolol in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: GZGD04112
Record Dates: First submitted 2012-08-06; First posted 2012-08-08 (Estimated); Last update posted 2015-03-23 (Estimated); Status verified 2015-03

CONDITIONS: Healthy
Keywords: Drug-drug interaction
MeSH Terms: interventions — eliglustat; Metoprolol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Metoprolol alone then eliglustat + metoprolol (Experimental): In Period 1 all participants will receive a single oral dose of metoprolol 50 mg on Day 1. In Period 2, participants will receive repeat oral doses of eliglustat 150 mg twice a day from Day 3 to Day 8 and a single oral dose of metoprolol 50 mg on Day 7.
  Interventions: Drug: Eliglustat; Drug: Metoprolol

INTERVENTIONS:
Drug: Eliglustat — Capsules for oral administration
  Other Names: Genz-112638
Drug: Metoprolol — Tablets for oral administration
  Other Names: Lopressor

SUMMARY:
The primary objective is to determine the effect of repeated oral doses of eliglustat 150 mg twice daily (BID) on the pharmacokinetics (PK) of orally administered metoprolol 50 mg in healthy adults.

The secondary objective is to assess the safety and tolerability of a single oral dose of metoprolol 50 mg when administered alone and in combination with repeated oral doses of eliglustat 150 mg BID in healthy adults.

ELIGIBILITY:
Inclusion Criteria:

1. The subject is willing and able to provide signed informed consent.
2. The male or female subject is in good general health and between 18 and 40 years of age, inclusive.
3. The subject has a body weight of 50 to 100 kg (110 to 220 lb) with a body mass index (BMI) ≤32 kg/m2 at screening.
4. The subject's physical examination, laboratory, vital sign, and electrocardiogram (ECG) test results are within normal limits at screening and Day -1 or, if abnormal, are not considered clinically significant in the opinion of the Investigator.
5. The subject has been a non-smoker for at least 6 months prior to the time of providing informed consent, and is willing and able to abstain from smoking (and use of other forms of nicotine) until completion of the safety follow-up visit.
6. The subject has not used drugs of abuse for at least 6 months prior to Day -1 and is willing and able to abstain from using drugs of abuse until completion of the safety follow-up visit.
7. The subject is willing and able to abstain from alcohol for 48 hours prior to the first dose of study drug until completion of the safety follow-up visit.
8. The subject is willing and able to abstain from grapefruit, grapefruit juice or any other grapefruit-containing products for 72 hours prior to the first dose of study drug until completion of the safety follow-up visit.
9. The subject is willing and able to maintain a normal-fiber diet (i.e., to abstain from excess fiber-rich foods) for 72 hours prior to the first dose of study drug until completion of the safety follow-up visit.
10. Female subjects of childbearing potential must have a documented negative pregnancy test at screening, Day -1 and prior to dosing on Day 7 and be willing to use a medically accepted form of contraception (as defined in the protocol) from screening until 30 days after the last dose of study drug. A woman of childbearing potential is defined as any female who has not been amenorrheic for at least 2 years or has not undergone a hysterectomy or surgical sterilization.

Exclusion Criteria:

1. The subject is classified as a cytochrome P450 2D6 (CYP2D6) poor metabolizer (or an indeterminate metabolizer with neither allele known to be active) based on results of CYP2D6 genotyping performed at screening. (Note: Prior CYP2D6 genotyping results may be used for the purpose of determining study eligibility if a copy of the laboratory report is available and the genotyping results can be interpreted with the same classification system used by the study reference laboratory.)
2. The subject has a digestive disorder, including malabsorption, gastroenteritis, pancreatitis, gastroesophageal reflux disease, inflammatory bowel disease (including Crohn's disease), or any other digestive disorder which, in the opinion of the Investigator, may affect oral bioavailability (e.g., clinically significant constipation, diverticulitis, or irritable bowel syndrome).
3. The subject has had a gastrointestinal (GI) surgical procedure that might affect drug transit time, (e.g., cholecystectomy, GI bypass surgery, partial or total gastrectomy, or small bowel resection).
4. The subject has any of the following: Clinically significant coronary artery disease including history of myocardial infarction or ongoing signs or symptoms consistent with cardiac ischemia or heart failure; clinically significant arrhythmias or conduction defect such as 2nd or 3rd degree atrioventricular (AV) block, a PR interval ≥200 msec, complete bundle branch block, prolonged QTc interval (e.g., repeated demonstration of a QTc interval ≥430 msec for male subjects and ≥450 msec for female subjects), sustained ventricular tachycardia, heart rate <55 beats/min, or systolic blood pressure <110 mmHg.
5. The subject has a clinically significant organic disease, including cardiovascular, renal, hepatic, gastrointestinal, pulmonary, neurologic, endocrine, metabolic, or psychiatric disease, or other medical condition, serious intercurrent illness, or extenuating circumstance that, in the opinion of the Investigator, precludes participation in the trial.
6. The subject has a disease, clinical finding, or any contraindication that would prohibit the use of metoprolol in a phase 1 study (i.e., risk of disease exacerbation outweighs benefit). Examples of these are clinical findings of glucose intolerance, poor arterial peripheral circulation or bronchospastic disease including asthma.
7. The subject has a history of fainting, postural lightheadedness, or any other postural symptoms.
8. The subject has received any prescription or non-prescription medication (with the exception of nonprescription-strength ibuprofen and acetaminophen, topical non-steroidal preparations, and topical hydrocortisone (up to 1% strength)) or dietary or herbal or fiber supplement within 30 days or 5 half-lives (whichever is longer) prior to the first dose of study drug without the approval of both the Investigator and Sponsor.
9. The subject has received an immunization within 30 days of providing informed consent.
10. The subject has received an investigational product within 30 days prior to the first dose of study drug or plans to receive any other investigational product at any time during the course of this study.
11. The subject has a history of drug allergies that are clinically significant in the opinion of the Investigator (e.g., significant rash or hives).
12. The subject has a screening laboratory test result above the upper limit of normal for any of the following liver function tests: aspartate aminotransferase (AST), alanine aminotransferase (ALT), gamma glutamyltransferase (GGT), and total bilirubin.
13. The subject tests positive for human immunodeficiency virus (HIV) antibody, hepatitis C antibody, or hepatitis B surface antigen at screening.
14. The subject tests positive for urine drugs of abuse, urine alcohol, or urine cotinine at screening.
15. The subject donated blood or blood products within 30 days prior to providing informed consent.
16. The subject's schedule or travel plans prevent the completion of all required visits.
17. The subject is scheduled for inpatient hospitalization, including elective surgery (inpatient or outpatient), during the study.
18. The subject has a history of cancer, with the exception of basal cell carcinoma.
19. The female subject of childbearing potential is pregnant or lactating.
20. The subject, in the opinion of the Investigator, is unable to adhere to the requirements of the study.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2012-05; Primary Completion 2012-06 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Metoprolol area under the plasma concentration time curve from time zero to the last evaluable concentration (AUC0-last) | Day 1 and Day 7; predose and up to 48 hours after drug administration
Metoprolol area under the plasma concentration time curve from time zero extrapolated to infinity (AUC0-∞) | Day 1 and Day 7; Predose and up to 48 hours after drug administration

SECONDARY OUTCOMES:
Maximum plasma concentration (Cmax) for metoprolol | Day 1 and Day 7; Predose and up to 48 hours after drug administration
Time to maximum plasma concentration (Tmax) for metoprolol | Day 1 and Day 7; Predose and up to 48 hours after drug administration
Terminal elimination half-life (T1/2) for metoprolol | Day 1 and Day 7; Predose and up to 48 hours after drug administration
Trough plasma concentration of eliglustat | Day 3, Day 4, Day 5, Day 6, Day 7 and Day 8.
  Eliglustat plasma concentration observed just prior to administration during repeated dosing.
Maximum plasma concentration (Cmax) of eliglustat | Day 7, up to 12 hours after drug administration
Time to maximum plasma concentration (Tmax) of eliglustat | Day 7; up to 12 hours after drug administration
Eliglustat area under the plasma concentration time curve during the dosing interval (AUC0-τ) | Day 7; up to 12 hours after drug administration
Number of participants with adverse events | Day 1 through to Day 14

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Genzyme, a Sanofi Company
Locations (1):
- Austin, Texas, United States